CLINICAL TRIAL: NCT05268653
Title: Investigation of the Effect of Motivational Interviewing on Obese Adolescents on Anthropometric Results, Nutrition, Exercise Behavior and Sedentary Activity Level
Brief Title: Motivational Interviewing Nutrition Exercise Obese Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Hasan EVCİMEN, Lecturer, Muş Alparslan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12.01.2021/1-1
Record Dates: First submitted 2022-01-11; First posted 2022-03-07 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Adolescent Obesity
Keywords: obesıty; motivational interviewing; sedentary actıvıty; nutrıtıon; exercıse
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled study in a quasi-experimental design in the pre-test post-test design.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational İnterviewing Group (Experimental): For the Motivational Interviewing (MI) treatment group, a clinical public health nursing doctoral student trained in Motivational Interviewing administered six motivational interviewing therapy sessions, each 30 minutes long. A 3-month follow-up will then be applied.
  Interventions: Behavioral: Motivatıonal İnterviewing (Treatment Group)
- Control Group (No Intervention): No attempt will be made

INTERVENTIONS:
Behavioral: Motivatıonal İnterviewing (Treatment Group) — Obese adolescents will be given a 6-session motivational interview.
  Arms: Motivational İnterviewing Group

SUMMARY:
This study is a randomized controlled study in a quasi-experimental design in the pre-test post-test design.The aim of this study is to examine the effect of motivational interview applied to obese adolescents on nutritional exercise behavior, anthropometric measurements and sedentary activity level.The data of this study were collected using a personal information form, Nutrition exercise behavior scale, Adolescent Sedentary Activity Questionnaire and anthropometric measurement form.In this study, nursing initiatives include a MG-based training program that will be given to obese adolescents in the experimental group in the form of 6 sessions after collecting preliminary test data. The final tests will be collected after 3 months of follow-up. Pre-test and post-test will be applied to the adolescents in the control group. Each training will take 30 minutes. Various training methods and techniques such as oral expression, question and answer, brainstorming, feedback and powerpoint presentations will be used within the scope of the training program

DETAILED DESCRIPTION:
Obesity has been increasing in children and adolescents as well as adults in recent years. Many factors play a role in the formation of obesity. The most important of these are sedentary lifestyle, wrong diet and insufficient physical activity. Motivational interviewing technique seems to give promising results in order to change risky health behaviors that cause obesity in adolescents. This study is a randomized controlled study in a quasi-experimental design in the pre-test post-test design.The aim of this study is to examine the effect of motivational interview applied to obese adolescents on nutritional exercise behavior, anthropometric measurements and sedentary activity level.The data of this study were collected using a personal information form, Nutrition exercise behavior scale, Adolescent Sedentary Activity Questionnaire and anthropometric measurement form.In this study, nursing initiatives include a MG-based training program that will be given to obese adolescents in the experimental group in the form of 6 sessions after collecting preliminary test data. The final tests will be collected after 3 months of follow-up. Pre-test and post-test will be applied to the adolescents in the control group. Each training will take 30 minutes. Various training methods and techniques such as oral expression, question and answer, brainstorming, feedback and powerpoint presentations will be used within the scope of the training program.

ELIGIBILITY:
Inclusion Criteria:

* being above the 95th percentile
* not going to a dietitian

Exclusion Criteria:

* having mental health problems

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Change in nutrition and exercise behavior scale score | baseline to 3 months
  The Nutrition and Exercise Behavior Scale (NEBS) is a five-point Likert-type scale consisting of 45 items and four sub-factors. Scale scores are evaluated in line with the scores obtained from the scale sub-dimensions. The score distribution of "Psychological/addictive eating behavior sub-factor" is between 11-55. A high score indicates psychological/addictive eating behavior. The score distribution of "Healthy nutrition-exercise behavior sub-factor" is between 14-70. A high score indicates healthy eating and exercise behavior. The score distribution of "unhealthy nutrition exercise behavior sub-factor" is between 14-70. A high score indicates unhealthy eating and exercise behavior. The "meal order sub-factor" score distribution is between 6-30. A high score indicates good meal order.
Change in adolescent sedentary actıvıty time | baseline to 3 months
  The original Adolescent Sedentary Actıvıty Questionnaire (ASAQ) has 11 questions for weekdays and 12 questions for weekends. ASAAQ covers pre-school and after-school time for each weekday, and all hours of the day for weekend days. The ASAA adapted into Turkish includes the time spent for 10 different SAs. Thus, the time spent for sedentary activities all week, weekdays and weekends can be calculated. In this context, the time spent in each activity category can be calculated. With ASAQ, sedentary activity times can be calculated for weekdays, weekends and the whole week in five sedentary activity categories.

CONTACTS AND LOCATIONS:
Locations (1):
- Mus AlparlanU, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Evcimen H, Bilgin S. The Effect of Motivational Interview-Based Education on Nutrition Exercise Behavior, Sedentary Activity Duration, and Anthropometric Outcomes in Obese Adolescents. Public Health Nurs. 2025 Mar-Apr;42(2):930-939. doi: 10.1111/phn.13530. Epub 2025 Jan 2. PMID 39748503